CLINICAL TRIAL: NCT02521818
Title: Feasibility and Efficacy of Dietary Interventions for Cognitive Impairment in Older Adults
Brief Title: Dietary Treatments for Cognitive Impairment in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00066092
Record Dates: First submitted 2015-08-10; First posted 2015-08-13 (Estimated); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Mild Cognitive Impairment; Probable Alzheimer's Disease
Keywords: cognition; dementia; neuropsychological; elderly; nutrition; diet
MeSH Terms: conditions — Cognitive Dysfunction; Dementia | interventions — Diet, Ketogenic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Modified Atkins Diet (Experimental): modified Atkins diet; fewer than 20 mg. carbohydrates per day, supplemented by extra dietary fats
  Interventions: Other: Modified Atkins Diet
- NIA Diet for Seniors (Active Comparator): Diet recommended by NIA for seniors
  Interventions: Other: NIA Diet for Seniors

INTERVENTIONS:
Other: Modified Atkins Diet
  Other Names: ketogenic diet
  Arms: Modified Atkins Diet
Other: NIA Diet for Seniors
  Arms: NIA Diet for Seniors

SUMMARY:
This trial seeks to establish the feasibility of implementing a ketogenic, modified Atkins diet (MAD) to older adults with mild cognitive impairment (MCI) or early Alzheimer's disease (AD) living in the community. A secondary aim is to determine whether adherence to the MAD results in better cognitive test scores than adherence to a non-ketogenic control diet. A final aim is to determine the role of apolipoprotein E (ApoE) genotype in participants' response to the MAD. Participants will be randomly assigned to a 12-week trial of either the MAD or a placebo diet based on the National Institute on Aging's recommendations for senior nutrition.

DETAILED DESCRIPTION:
It is well established that Alzheimer's disease (AD) is associated with insulin resistance and, hence, abnormal glucose metabolism. In fact, abnormalities in the brain's uptake of glucose can be observed on PET imaging in advance of clinical symptoms. In patients with established dementia due to AD, the severity of cognitive impairment is strongly correlated with the decrease in glucose uptake. Ketone bodies, the products of fat metabolism, can serve as a "backup" fuel when glucose is unavailable. Ketone body metabolism appears to bypass the metabolic processes that are abnormal in AD and may provide better nourishment for neurons. As a result, ketone body metabolism may slow cognitive decline or even improve cognition in patients with AD.

Participants will be 60 people, age 60 or older, with MCI or mild probable AD and without significant cardiovascular disease. They will be required to obtain the consent of their primary care physicians for their participation. Each patient will have a study partner who is cognitively healthy, lives with the participant, and can help him/her adhere to the diet. A research dietitian will teach participants and partners the new diet and monitor participants' adherence with food logs, in-person assessments, and urine ketone testing. After an initial baseline visit, participants will complete four in-person assessments during which adherence to the diet will be assessed and neurocognitive tests will be administered. It is hypothesized that the MAD will be feasible and well tolerated by seniors with MCI and AD. It is further hypothesized that adherence to the MAD will be associated with a greater increase (or less decline) in cognitive test scores than the placebo diet, particularly for those participants who do not carry an ApoE ε4 allele.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of mild cognitive impairment or Alzheimer's disease
* availability of cohabitating study partner without cognitive impairment
* consent of primary care physician

Exclusion Criteria:

* history of stroke
* history of coronary artery disease
* history of pancreatitis
* untreated hypothyroidism or B12 deficiency
* history of renal disease or recurrent kidney stones
* history of liver disease
* insulin-dependent diabetes
* body mass index <18.5
* multiple food allergies
* follow strict diet (e.g., vegetarian, gluten-free)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Feasibility for MAD Group | 12 weeks
  Achieving moderate ketosis (>=40 mg.dl) at 3 consecutive follow-up visits
Feasibility for Control Group | 12 weeks
  Achieving a Healthy Eating Index (>=85) at 3 consecutive follow-up visits

SECONDARY OUTCOMES:
Efficacy for Cognition | 12 weeks
  Composite Memory Score (mean z-score on delayed recall of HVLT-R and BVMT-R)
Efficacy for Function | 12 weeks
  Change in MDS-HC Instrumental Activities of Daily Living Score

CONTACTS AND LOCATIONS:
Overall Officials: Jason Brandt, Ph.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States